CLINICAL TRIAL: NCT07015879
Title: Evaluation of the Effect of Continuous Care Counseling Based on Roy's Adaptation Model on Comfort and Quality of Life in Patients Undergoing Total Knee Arthroplasty: A Randomized Controlled Trial
Brief Title: The Effect of Continuous Care Counseling Based on the Roy Adaptation Model on Comfort and Quality of Life in Patients Undergoing Total Knee Arthroplasty
Acronym: RAM-TKA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cyprus International University (Other)
Responsible Party: Principal Investigator, Prof. Dr. Sıddıka Fatma Uygur, prof. dr., Cyprus International University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TDP-RAM-
Record Dates: First submitted 2025-06-03; First posted 2025-06-11 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: Osteoarthritis; Care Model; Quality of Life; Nursing Interventions; Knee
Keywords: Knee osteoarthritis; Total knee arthroplasty; Roy Adaptation Model; Continuous care; Comfort; Quality of life; Nursing; Postoperative care; Patient education
MeSH Terms: conditions — Osteoarthritis; Osteoarthritis, Knee

STUDY DESIGN:
Intervention Model Description: Participants were randomly assigned to either the intervention group, which received continuous care counseling based on the Roy Adaptation Model, or the control group, which received standard postoperative care. Data were collected preoperatively, on the second postoperative day, and at the first and third months after discharge.
Masking Description: This study is an open-label study. Due to the nature of continuous care counseling, it is not possible for participants and care providers to be unaware of the intervention
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Continuous Care Counseling Based on the Roy Adaptation Model (Experimental): Patients in the experimental group will receive video-supported education with verbal explanation in the clinic five days before surgery; the session will be repeated one day before surgery to assess patient comprehension. The instructional video will remain accessible to the patient, and home-care precautions will be reviewed at discharge. Overall comfort and quality of life will be measured face-to-face both before and after surgery, and by telephone at the first and third months following discharge. Adherence to watching the video, performing prescribed exercises, and any postoperative complications will also be monitored.
  Interventions: Behavioral: Continuous Care Counseling Based on the Roy Adaptation Model
- Control Group (No Intervention): Patients will receive the clinic's routine treatment and nursing care.

INTERVENTIONS:
Behavioral: Continuous Care Counseling Based on the Roy Adaptation Model — Patients in the control group will receive the clinic's routine treatment and nursing care. This care includes preoperative and postoperative information, prevention of leg flexion, monitoring of vital signs, pain management, discharge education, and discharge of patients without complications three days after surgery. In addition, patients' overall comfort and quality of life will be assessed face-to-face five days before surgery and on the second postoperative day, and by telephone at the first and third months after discharge.
  Arms: Continuous Care Counseling Based on the Roy Adaptation Model

SUMMARY:
Osteoarthritis is a common joint disease that leads to problems such as pain, restricted mobility, and decreased quality of life in the knee joint, especially among elderly individuals. In advanced-stage knee osteoarthritis, total knee arthroplasty (TKA) is performed to reduce pain and loss of function. However, in the postoperative period, patients may encounter various problems such as pain, sleep disturbances, anxiety, and difficulties in daily living activities.

This study investigates how continuous care counseling based on Roy's Adaptation Model affects the comfort and quality of life of patients undergoing total knee arthroplasty. Roy's Adaptation Model is a widely used approach in nursing that supports individuals in adapting to changes they experience. Counseling and education provided in line with this model aim to help patients cope with the physical and psychological problems they face before and after surgery.

In the study, specially designed training and counseling services were offered to patients who underwent surgery, and the effects of these services on pain, anxiety, sleep quality, and daily living activities were evaluated. The results of the research indicate that continuous care counseling based on Roy's Adaptation Model may be effective in improving patients' postoperative comfort and quality of life. These findings may contribute to the improvement of postoperative care for both patients and healthcare professionals.

DETAILED DESCRIPTION:
Osteoarthritis is a chronic joint disease that affects millions of people worldwide and is particularly prevalent among the elderly population. Knee osteoarthritis leads to significant problems such as severe pain, restricted mobility, and loss of independence, thereby negatively impacting quality of life. In advanced stages of knee osteoarthritis, total knee arthroplasty (TKA) is a commonly preferred surgical method to reduce pain and loss of function. However, in the postoperative period following TKA, patients may experience multidimensional problems such as pain, sleep disturbances, psychological stress, anxiety, and difficulties in daily living activities.

In modern nursing practice, the management of these problems experienced by patients before and after surgery and the improvement of their quality of life are of great importance. Roy's Adaptation Model is a theoretical framework frequently utilized in nursing that supports individuals in adapting to environmental changes and stressors. This model advocates for a holistic assessment of patients in terms of their physiological, psychological, social, and role functions, and for the structuring of care plans accordingly.

This study aims to evaluate the effect of continuous care counseling based on Roy's Adaptation Model on the comfort and quality of life of patients undergoing total knee arthroplasty. In the research, specially designed training and counseling services were provided to patients who underwent surgery, and the effects of these services on pain, anxiety, sleep quality, and daily living activities were evaluated using both quantitative and qualitative methods. Within the scope of the study, patients in the intervention group received continuous care counseling and video-supported education based on the Roy Adaptation Model, while the control group received standard care. Data were collected and analyzed using quality of life and comfort scales.

The findings of the study indicate that continuous care counseling based on Roy's Adaptation Model may be effective in improving postoperative comfort and quality of life in patients undergoing total knee arthroplasty. These results may contribute to the improvement of postoperative care and the development of patient-centered care practices for both patients and healthcare professionals.

ELIGIBILITY:
Inclusion Criteria:

Provided written and verbal consent to participate in the study Aged 18 years or older Conscious, oriented, and cooperative Able to speak and understand Turkish Has the ability to speak, hear, and see Has no diagnosed psychiatric illness Has no known cancer diagnosis Undergoing elective surgical intervention Undergoing total knee arthroplasty (TKA) for the first time Undergoing unilateral TKA

Exclusion Criteria:

Undergoing emergency surgical intervention Readmission for revision surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2024-06-23 (Actual); Primary Completion 2024-11-19 (Actual); Study Completion 2025-03-14 (Actual)

PRIMARY OUTCOMES:
Overall Comfort Level | Preoperative (5 days before surgery), postoperative 2nd day, and at the 1st and 3rd months after discharge
  Patients' overall comfort levels will be assessed using the "General Comfort Questionnaire Short Form" 5 days before surgery, on the 2nd day after surgery, and at the 1st and 3rd months after discharge.

SECONDARY OUTCOMES:
Overall Quality of Life | Preoperative (5 days before surgery), postoperative 2nd day, and at the 1st and 3rd months after discharge
  Patients' quality of life will be measured using the "General Quality of Life Scale" at the same time points (preoperative, postoperative day 2, 1st and 3rd months after discharge).

CONTACTS AND LOCATIONS:
Overall Officials: Burcu Dikmen, PhD, Principal Investigator — Cyprus International University
Locations (1):
- Cyprus International University, Mersin, Lefkosa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No